CLINICAL TRIAL: NCT00660270
Title: A Phase II Trial Of Adjuvant Chemoradiation Following Pancreatic Resection For Adenocarcinomas Of The Pancreas Using 3-D Conformal Radiation With Cisplatin, 5FU, And Alpha-Interferon As Radiosensitizing Agents Followed By Gemcitabine
Brief Title: Chemotherapy and Radiation Following Pancreatic Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-0307
Record Dates: First submitted 2008-04-11; First posted 2008-04-17 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Pancreatic Cancer
Keywords: Chemotherapy; Radiation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiotherapy; Cisplatin; Fluorouracil; Interferon-alpha; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Surgery (pancreaticoduodenectomy, either standard or pylorus-preserving, with either standard or extended lymph node dissection, with or without portal vein resection) should occur at 8 weeks (plus or minus 2, not to exceed 10)
  Radiation therapy will occur 8 weeks (plus or minus 2, not to exceed 10) postoperatively. Daily dose of 1.8 Gy five days per week. The first 45 Gy will be given to planning target volume 1. After 45 Gy, portals will be reduced to encompass planning target volume 2. The boost dose will be 5.4 Gy.
  Cisplatin IV 25 mg/m2 on days 1, 8, 15, 22, 29, and 36 during radiation.
  5-FU CIVI at 175 mg/m2/d on days 1-38 without interruption during radiation.
  Alpha-interferon SQ 3,000,000 units on Mondays, Wednesdays, and Fridays during radiation therapy.
  Gemcitabine IV 1000 mg/m2 4 weeks after conclusion of radiation (on a 3 weeks on/1 week off schedule) on days 71, 78, 85, 99, 106, and 113.
  Interventions: Procedure: Pancreatic Surgery; Radiation: Radiation therapy; Drug: Cisplatin; Drug: 5-FU; Drug: Alpha-interferon; Drug: Gemcitabine

INTERVENTIONS:
Procedure: Pancreatic Surgery
Radiation: Radiation therapy
Drug: Cisplatin
  Other Names: CDDP; Platin
Drug: 5-FU
  Other Names: Fluorouracil; Efudex
Drug: Alpha-interferon
Drug: Gemcitabine
  Other Names: Gemzar

SUMMARY:
To describe the overall survival and disease-free survival in pancreatic cancer patients treated with adjuvant chemoradiation with cisplatin, continuous infusion 5FU and interferon alpha followed by gemcitabine.

To describe the toxicities associated with adjuvant chemoradiation with cisplatin. 5FU and interferon alfa followed by gemcitabine in patients with pancreatic cancers.

DETAILED DESCRIPTION:
The adjuvant therapy of pancreas cancer has remained a challenge for oncology specialists from all disciplines since the initial development of the pancreaticoduodenectomy by Whipple in 1935 (Whipple, Ann Surg, 1935). A variety of phase II experiences utilizing radiation therapy and 5FU-based chemotherapy following curative surgery for pancreas cancer have consistently produced the disappointing survival results of 18-24 months median survival, 40%-50% 2-year survival and 10%-20% 5-year survival (Evans, in DeVita, et.al Cancer Principles and Practices of Oncology, 1997). Indeed, whether any adjuvant therapy following pancreaticoduodenectomy for pancreas cancer is of benefit to patients remains a debated question. The landmark study performed by the GITSG in patients with pancreatic cancer displayed a survival advantage for patients receiving postoperative radiation therapy and 5FU compared to those receiving pancreaticoduodenectomy only (2-year survival 43% vs. 18%, p=0.03). As a result, this study became to some the standard of care for patients with resected pancreas cancer in the US (GITSG, Cancer 1987). However, this study rightfully has been criticized from a variety of perspectives over the years; furthermore, recent experiences by the EROTC and ESPAC have failed to reproduce the GITSG results (Klinkenbijl, Ann Surg 1999,Neoptolemos, Proc ASCO 2000). However, the results of these two studies have also received significant criticisms. The EORTC data are underpowered and the study failed to use post-radiation chemotherapy to optimum advantage. The ESPAC data have been criticized as being statistically invalid by trial desig10/14/02n and analysis. Thus, the optimization of adjuvant therapy following pancreaticoduodenectomy for pancreas cancer remains a subject of debate and poses essentially the same challenge to oncology specialists at the beginning of the 21st century as it has for the past sixty years.

Confronted with these issues, investigators at the Virginia Mason Clinic began in 1995 a phase II trial utilizing cisplatin and alpha-interferon in conjunction with 5FU and radiation therapy following pancreaticoduodenectomy for pancreatic adenocarcinoma. The logic behind this protocol was as follows:

1. Recurrence following surgery and adjuvant chemoradiation in protocols for resected pancreas cancer to that date had been associated with a high incidence of both local and systemic recurrence; thus treatment must focus on improvement in relapse rates in both areas.
2. No chemotherapy regimens (as of 1995), either single agent or multi-agent, had shown response rates markedly different from that seen with single agent 5FU (typically on the order of 10%)
3. Therapeutic advance in the adjuvant therapy of pancreas cancer must therefore focus on systemic agents that have the potential to synergize the tumoricidal activity of radiation therapy and/or each other.
4. Cisplatin and alpha-interferon, like 5FU, do have radiosensitizing activity in experimental tumor systems and thus potentially could be added to 5FU to create a "combination" radiosensitizing agent analogous to the way chemotherapy agents are combined for systemic effect.
5. These chemotherapeutic agents also have direct synergistic anticancer activity with respect to each other in experimental tumor systems .
6. These agents also have, to a large extent, non-overlapping toxicities and can be delivered on an outpatient basis.

Using the above logic, a novel phase II protocol (with radiation therapy) for the adjuvant therapy of pancreas cancer was developed. The protocol was constructed as follows:

* XRT 5000cGy/200cGy fractions given daily M-F wks 1-5
* CDDP 30 mg/m2 d 1 wks 1-5
* IFN-A 3,000,000U sq qod wks 1-5 beginning d 1
* 5FU 200mg/m2 wks 1-5 beginning d 1; repeated wks 10-15 and wks 18-23 (2 6 wk chemotherapy courses post chemoradiation ).

Patients, in general, were treated within 8 weeks following pancreaticoduodenectomy (in general, performed as a pylorus preserving procedure without extended lymph node dissection) and included patients with adenocarcinomas of the head, body and tail of the pancreas. Other periampullary cancers were not included in this study.

The phase II trial from Virginia Mason has been published in a variety of forms, both abstract (Picozzi, Proc ASCO 1999,2000) and manuscript (Nukui, Am J Surg 2000). To date, 38 patients have been treated at Virginia Mason using this method. Average patient age is 64. Thirty three patients had cancers of the pancreas head, 5 patients had body and/or tail cancers. Noteworthy in this series is a particularly high incidence of the adverse disease prognostic factors for recurrence such as nodal involvement (79%) and non-surgical margin positivity (32%). Using a prognostic model for disease recurrence developed at Johns Hopkins incorporating the above factors plus tumor type (pancreatic head versus other periampullary cancers), tumor size, tumor differentiation and estimated blood loss at surgery, 37/38 patients (97%) were judged to be at high risk for disease recurrence.

Results of this trial updated as of February, 2001include the following important results:

* All patients (38/38) treated to date have completed the chemoradiation phase of treatment (wks 1-5); 35/38 patients completed the entire treatment course.
* Approximately 90% of planned chemotherapy was delivered; virtually all planned radiation therapy was delivered.
* Toxicity has been almost entirely GI-related (anorexia/dehydration, mucositis, nausea/vomiting, diarrhea).
* As a result of the above toxicity, the majority of patients required treatment delays during chemoradiation and approximately 30% (13/38) required hospitalization. However, there have been no treatment-related fatalities, and all patients have regained full functional status.
* Median follow-up at present is greater than 2 years; 21/38 patients have been followed for greater than 2 years. 28/38 (74%) patients remain alive, and 25/38 (67%) patients remain alive and disease free.
* At present, the median survivorship of this patient cohort is in excess of 45 months (45.8 months, 95% confidence limits 36-55 months); the actuarial 2-year and 5-year survivorships are 65 % and 60 %, respectively. 13/21 patients followed for more than two years remain alive at this time (including 3 patients alive more than 5 years from initial diagnosis). If just the 33 patients with adenocarcinomas of the pancreas head in this phase II trial are considered, the median survivorship rises to 49 months (95% confidence limits 39-59 months). Actuarial 2-year and 5-year survivorships are 73% and 68% respectively.
* All recurrences have taken place between 5 and 22 months from the time of diagnosis (none later).
* The recurrence pattern seen to date is as follows; 2 patients local recurrence, 7 patients systemic and 4 patients both local and systemic recurrence. The local control rate has thus been approximately 85% (32/38 patients) and the systemic control rate approximately 70% (27/38 patients).

More detailed data on all 38 patients with adenocarcinomas of the pancreas treated using this protocol at Virginia Mason to date are displayed in Figure 1.

These data were presented to the Pancreas Cancer Committee of the ACOSOG in December,2000. Meeting participants agreed to further development of this protocol given the treatment results seen in comparison with the historical precedents previously cited. These outcomes were seen as particularly favorable given the high-risk nature of the patient population studied. However, the protocol also received the following criticisms from meeting participants, including NCI reviewers. First, the protocol had only been studies to date at a single institution. Second, the toxicity of the regimen was seen as quite significant, especially during chemoradiation, when 30% of patients were hospitalized. Finally, the post-chemoradiation phase of chemotherapy (infusional 5FU only) was seen as potentially suboptimal, as several types of chemotherapy regimens, including both combination regimens utilizing infusional 5FU(ref) and gemcitabine (ref) have produced superior response rates in phase II trials to that seen with single agent 5FU. As a result of the above dialog, it was decided by the ACOSOG Pancreas Cancer committee to develop a multi-institutional phase II trial based upon the Virginia Mason protocol that would incorporate the above comments. It was also felt that this effort should not conflict with a phase III protocol being planned by the committee comparing a multi-agent 5FU-based regimen developed at UCLA with radiation therapy with the single agent 5FU approach used by the GITSG.

To address the protocol-related concerns mentioned above, the following modifications in the original Virginia Mason protocol are suggested:

The issue of toxicity during chemoradiation is addressed in three ways. First, radiation therapy will be delivered to more confined fields, particularly given the predominance of systemic recurrence in the therapeutic results to date. Second, the dose intensity of the chemotherapy agents (cisplatin, 5FU, Alpha-interferon) given during radiation will be reduced slightly. This is done remembering the majority of patients (approximately 70%) did require a break in treatment during this phase of therapy. Finally, to assist other providers new to this protocol, a supportive care pathway has been developed to assist in avoidance of treatment related toxicity (e.g. nausea, gastritis, hyperglycemia) during treatment.

ELIGIBILITY:
* Resected adenocarcinoma of the pancreas
* ECOG performance status 0 or 1
* No prior chemotherapy or radiation therapy for cancer within the last five years.
* Prior history of other malignancies allowable, if stable or requiring no active therapy.
* Absolute neutrophil count >/= 1,500/mm3, platelet count >/= 100,000/mm3, and hemoglobin >/= 9 g/dL.
* Serum creatinine </= 2 mg/dL.
* Serum bilirubin </= 3.0 mg/dL.
* Serum transaminases ( SGOT and SGPT) </= 5-fold the institutional upper limits.
* No co-existing severe medical illnesses, such as unstable angina, uncontrolled diabetes mellitus, uncontrolled arrhythmia or uncontrolled infection.
* Able to sign an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2002-05; Primary Completion 2006-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To describe the overall survival and disease-free survival | 2 years

SECONDARY OUTCOMES:
To describe the toxicities associated with adjuvant chemoradiation with cisplatin, 5FU and interferon alfa followed by gemcitabine in patients with pancreatic cancers. | Week 15

CONTACTS AND LOCATIONS:
Overall Officials: David Linehan, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Linehan DC, Tan MC, Strasberg SM, Drebin JA, Hawkins WG, Picus J, Myerson RJ, Malyapa RS, Hull M, Trinkaus K, Tan BR Jr. Adjuvant interferon-based chemoradiation followed by gemcitabine for resected pancreatic adenocarcinoma: a single-institution phase II study. Ann Surg. 2008 Aug;248(2):145-51. doi: 10.1097/SLA.0b013e318181e4e9. PMID 18650621
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu